CLINICAL TRIAL: NCT02672631
Title: Evaluation of Primary Repaired Wrist Level Complete Median Nerve Transection With Clinical, Electroneuromyographic (ENMG) and Diffusion Tensor Imaging (DTI) Methods
Brief Title: Evaluation of Complete Median Nerve Transection With Clinical, Electroneuromyographic and Diffusion Tensor Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, İbrahim Karaman, assistant professor doctor, TC Erciyes University
Other Study IDs: ENMG and MRI on Median Nerve
Record Dates: First submitted 2016-01-19; First posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Wound, Healed (Morphologic Abnormality); Injury of Median Nerve
MeSH Terms: conditions — Wounds and Injuries | interventions — Restraint, Physical; Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Median Nerve injury hand: Participants will be randomly called; and that 10 participants which had unilateral median nerve transection totally and repaired primely in our clinic at 2014. In the sample, correlations between physical examination (Tinnel Test, motor strength assessment (Medical Research Council (MRC) Scale), static two-point discrimination test (S2PD), Semmes-Weinstein (SW) monofilament test, the Disability of the Arm, Shoulder and Hand (DASH) test), ENMG with the DTI results will be assessed.
  Interventions: Other: physical examination; Other: DTI; Other: ENMG
- Healthy Hand: Control group will be taken from patients other hand which had not injured before. And we will compare with first group's results.
  Interventions: Other: physical examination; Other: DTI; Other: ENMG

INTERVENTIONS:
Other: physical examination — Investigators will apply for evaluate clinical median nerve function to all of groups. (Adductor pollicis power (x/5), sense exam(normal/hipoestesia/anestesia) of hand, tinnel test(+/-), DASH score, DN4 neuropathic pain score)
Other: DTI — Investigators will apply for evaluate median nerve healing countable results to all of groups (apparent diffusion coefficient for avarage diffusion (ADC) and fractional anisotropy diffusion orientation(FA) - FA :0 means diffusion is homogenic FA:1 means tissue has heterogenic diffusion
  Other Names: Diffusion Tensor Imaging
Other: ENMG — Investigators will apply for evaluate median nerve healing countable results to all of groups. And they will evaluate motor nerve transmission speed, sensitive nerve transmission speed and united muscle action potential
  Other Names: Electroneuromyography

SUMMARY:
The aim of this study is to determine whether clinical, sensory and motor development correlated with the values obtained from Electroneuromyography and DTI in postoperative follow up patients who underwent primary repair after the total median nerve injuries.

Median nerve is one of three major nerves of hand and forearm and often injure with glass etc, in follow up of healing; clinical examination and ENMG are often used. Both of these methods are subjective, noninvasive and objective new method is required. In this context; differences between intact, recovering and not healed nerve tissue's diffusions have led to the hypothesis; "The recovery of the repaired nerve tissue can be monitored by Diffusion Tensor Imaging method".

DETAILED DESCRIPTION:
The aim of this study is to determine whether clinical, sensory and motor development correlated with the values obtained from Electroneuromyography and DTI in postoperative follow up patients who underwent primary repair after the total median nerve injuries.

Median nerve is one of three major nerves of hand and forearm. It is below flexor tendon and retinaculum at the level of the wrist and often injured at this level and subtotally. The primary microsurgical suture technique under a microscope is the gold standard treatment. In follow up of healing; clinical examination and ENMG are often used. Both of these methods are subjective, although ENMG is more objective, however that is an invasive method, and need experienced neurologists. So, noninvasive and objective new method is required. In this context; differences between intact, recovering and not healed nerve tissue's diffusions have led to the hypothesis; "The recovery of the repaired nerve tissue can be monitored by Diffusion Tensor Imaging method". There is no similar study in the literature.

Ten patients who were operated for median nerve injuries in 2014 will be enrolled. In the sample, correlations between Tinnel Test, motor strength assessment (Medical Research Council (MRC) Scale), static two-point discrimination test (S2PD), Semmes-Weinstein (SW) monofilament test, the Disability of the Arm, Shoulder and Hand (DASH) test, EMG with the DTI results will be assessed.

At the end of the study; it is expected that a significant correlation between conventional methods and DTI. If the results support the hypothesis; DTI may get to the literature as noninvasive and objective method in follow of nerve regeneration.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 years old
* Total and isolated median nerve transection

Exclusion Criteria:

* Under 18 and over 40 years old
* Partially transection of median nerve
* Median nerve transection with radial or ulnar nerve injury

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Ten patients who were operated for median nerve injuries in 2014 will be enrolled. In the sample, correlations between Tinnel Test, motor strength assessment (Medical Research Council (MRC) Scale), static two-point discrimination test (S2PD), Semmes-Weinstein (SW) monofilament test, the Disability of the Arm, Shoulder and Hand (DASH) test, EMG with the DTI results will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Electroneuromyography | 2 months
  conventional evaluation of nerve healing - That evaluate axonal transfer speed etc
Physical Examination | 2 months
  conventional evaluation of nerve healing. That Evaluate sensitivity, motor functions and paresthesia

SECONDARY OUTCOMES:
Diffusion Tensor Imaging Methods | 2 months
  new method for evaluation of nerve healing with tissues diffusion on magnetic resonants imaging

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Karaman, ass.doc.dr, Study Director — TC Erciyes University
Locations (1):
- Erciyes University Faculty of Medicine, Melikgazi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Study Protocol — http://clinical-mri.com/mr-neurography-diagnostic-criteria-to-determine-lesions-of-peripheral-nerves/